CLINICAL TRIAL: NCT06472908
Title: Efficacy and Safety of Colchicine After Percutaneous Coronary Intervention
Brief Title: Efficacy and Safety of Colchicine After PCI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Director in the department of cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COLPCI
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Coronary Heart Disease; Percutaneous Coronary Intervention; Colchicine
MeSH Terms: conditions — Coronary Disease | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Colchicine 0.5 mg (Experimental): Colchicine 0.5 mg, one pill a day, oral intake
  Interventions: Drug: Colchicine 0.5 mg
- Colchicine 0.375 mg (Experimental): Colchicine 0.375 mg, one pill a day, oral intake
  Interventions: Drug: Colchicine 0.375 mg
- Placebo (Placebo Comparator): Placebo, one pill a day, oral intake
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 mg — Colchicine 0.5 mg, one pill a day, oral intake
  Other Names: no other name
  Arms: Colchicine 0.5 mg
Drug: Colchicine 0.375 mg — Colchicine 0.375 mg, one pill a day, oral intake
  Other Names: no other name
  Arms: Colchicine 0.375 mg
Drug: Placebo — Placebo, one pill a day, oral intake
  Other Names: no other name
  Arms: Placebo

SUMMARY:
Colchicine (0.5 mg/day) was recommended by the U.S. Food and Drug Administration in 2023 for the anti-inflammatory treatment of coronary heart disease (CHD). However, colchicine is still not approved for CHD treatment in China. There is no large-scale clinical evidence that colchicine can be used to treat Chinese patients with CHD. Considering the low body weight of the East Asian population, it is unclear whether the recommended standard dose (0.5 mg/day) is suitable for Chinese patients. Therefore, we need to further explore the effects of different doses of colchicine on the efficacy and safety of clinical endpoints in the Chinese population with CHD.

This study is a multicenter, prospective, randomized, controlled, double-blind, event-driven clinical study conducted in China. The primary objective of this study is to determine whether long-term treatment with different doses of colchicine reduces the incidence of cardiovascular events in Chinese patients undergoing PCI. The secondary objective is to determine the safety of long-term treatment with different doses of colchicine in this patient population.

DETAILED DESCRIPTION:
After informed consent, 8862 subjects who meet all inclusion will be randomly assigned to receive colchicine (0.5 mg/day), colchicine (0.375 mg/day), or placebo (1:1:1 allocation ratio), with follow-up at months (1, 6, 12, 18, 24…) after randomization, and phone assessments at months (3, 9, 15, 21…). The occurrence of any endpoints or other adverse events will be assessed every 3 months. Subjects will also receive standard medical care for antiplatelets, control of dyslipidemia, hypertension, angina and diabetes as directed by national guidelines. All suspected cardiovascular endpoints will be adjudicated by the Clinical Event Committee (CEC, consisting of three experienced members blinded as to allocation of therapy). The Data and Safety Monitoring Board (DSMB, consisting of five fully independent members) will review unblinded safety data as detailed in the DSMB charter. An interim analysis is planned after approximately 50% of primary endpoints have been positively adjudicated. The DSMB charter will pre-specify the methodology for the interim analysis and the rules for early termination of the study.

ELIGIBILITY:
Inclusion Criteria:

* (1) Capable and willing to provide informed consent;
* (2) Age ≥18 and ≤80 years old, regardless of sex;
* (3) Hospitalized patients with CHD requiring PCI;
* (4) Completion of all planned PCI during hospitalization;
* (5) Standardized treatment of coronary artery disease according to national guidelines.

Exclusion Criteria:

* (1) Known allergy to colchicine;
* (2) Colchicine taken within 10 days prior to randomization group;
* (3) Patients currently in cardiogenic shock or hemodynamically unstable;
* (4) Patients with known inflammatory bowel disease or chronic diarrhea;
* (5) Abnormal liver function (ALT> 3 times the upper limit of normal);
* (6) Abnormal renal function (eGFR<30mL/min/1.73m2);
* (7) Active malignant tumors reported in past medical history;
* (8) Existing or planned treatment with other anti-inflammatory or immunosuppressive drugs;
* (9) Pregnant women, lactating women or women of childbearing age who did not use effective contraceptives;
* (10) Any other circumstances in which the investigator judges that the patient is not suitable to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8862 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and ischemia-driven revascularization | An estimated 2-4 years period
  From randomization to the first occurrence

SECONDARY OUTCOMES:
Composite of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke | An estimated 2-4 years period
  From randomization to the first occurrence
Ischemia-driven revascularization | An estimated 2-4 years period
  The number of participants with Ischemia-driven revascularization
Nonfatal myocardial infarction | An estimated 2-4 years period
  The number of participants with myocardial infarction
Nonfatal stroke | An estimated 2-4 years period
  The number of participants with stroke
Urgent hospitalization for unstable angina | An estimated 2-4 years period
  The number of participants with urgent hospitalization for unstable angina
In-stent restenosis | An estimated 2-4 years period
  The number of participants with in-stent restenosis
Stent thrombosis | An estimated 2-4 years period
  The number of participants with stent thrombosis
Cardiovascular death | An estimated 2-4 years period
  The number of participants with cardiovascular death
All-cause mortality | An estimated 2-4 years period
  The number of participants with all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Cheng, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (36):
- China (36):
  - The Second Hospital & Clinical Medical School, Lanzhou University, Lanzhou, Gansu
  - Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The Central Hospital of Enshi Tujia and Miao Autonomous Prefecture, Enshi
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huangshi Central Hospital, Huangshi
  - Shandong Provincial Hospital, Jinan
  - Jingzhou Central Hospital, Jingzhou
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Songjiang Hospital Affiliated with Shanghai Jiao Tong University School of Medicine, Shanghai
  - The General Hospital of Northern Theater Command of the Chinese People's Liberation Army, Shenyang
  - Dongfeng General Hospital, Hubei University of Medicine, Shiyan
  - Shiyan Renmin Hospital, Shiyan
  - Taihe hospital, Shiyan
  - Suizhou Central Hospital, Suizhou
  - Shanxi Cardiovascular Disease Hospital, Taiyuan
  - China Resources and WISCO General Hospital, Wuhan
  - Fifth Hospital in Wuhan, Wuhan
  - Wuhan Asia Heart Hospital, Wuhan
  - Wuhan Central Hospital, Wuhan
  - Wuhan First Hospital, Wuhan
  - Wuhan Fourth Hospital, Wuhan
  - Wuhan Puren Hospital, Wuhan
  - Wuhan Sixth Hospital, Affiliated Hospital of Jianghan University, Wuhan
  - Wuhan Third Hospital, Wuhan
  - Wuhan Wuchang Hospital, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiangyang Central Hospital, Xiangyang
  - Xiangyang First People's Hospital, Xiangyang
  - Xianning Central Hospital, Xianning
  - Yichang Central People's Hospital, Yichang
  - Fuwai Huazhong Cardiovascular Hospital, Zhengzhou

REFERENCES:
- [Result] Lawler PR, Bhatt DL, Godoy LC, Luscher TF, Bonow RO, Verma S, Ridker PM. Targeting cardiovascular inflammation: next steps in clinical translation. Eur Heart J. 2021 Jan 1;42(1):113-131. doi: 10.1093/eurheartj/ehaa099. PMID 32176778
- [Result] Nelson K, Fuster V, Ridker PM. Low-Dose Colchicine for Secondary Prevention of Coronary Artery Disease: JACC Review Topic of the Week. J Am Coll Cardiol. 2023 Aug 15;82(7):648-660. doi: 10.1016/j.jacc.2023.05.055. PMID 37558377
- [Result] Fiolet ATL, Opstal TSJ, Mosterd A, Eikelboom JW, Jolly SS, Keech AC, Kelly P, Tong DC, Layland J, Nidorf SM, Thompson PL, Budgeon C, Tijssen JGP, Cornel JH. Efficacy and safety of low-dose colchicine in patients with coronary disease: a systematic review and meta-analysis of randomized trials. Eur Heart J. 2021 Jul 21;42(28):2765-2775. doi: 10.1093/eurheartj/ehab115. PMID 33769515